CLINICAL TRIAL: NCT03101202
Title: Comparison of Endotracheal Tube With Subglottic Suction Drainage With Standard Endotracheal Tube in the Incidence of Airway Colonization and Ventilator Associated Pneumonia
Brief Title: To Compare Endotracheal Tube (ET) With Subglottic Suction Drainage and Standard ET in the Incidence of VAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vijay Noel Nongpiur, Senior Resident, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IECPG-464/27.07.2016
Record Dates: First submitted 2017-03-24; First posted 2017-04-05 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Ventilator-Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SSD Arm (Experimental): In the SSD arm, the patients will be intubated with an endotracheal tube with suglottic suction drainage (SSD tube)
  Interventions: Device: SSD tube
- Standard Arm (No Intervention): In the standard arm, the patients will be intubated with the standard endotracheal tube which does not have subglottic suction.

INTERVENTIONS:
Device: SSD tube — The SSD tube allows the suction of subglottic secretions that collect above the cuff of the endotracheal tube
  Arms: SSD Arm

SUMMARY:
Ventilator Associated Pneumonia (VAP) is associated with increased hospitalisation, increased health care cost and high morbidity and mortality. The incidence of VAP increases with duration of mechanical ventilation. There is limited data especially from India on the incidence of VAP and also the role of subglottic aspiration in its prevention. The aim of this study is to determine the role of subglottic suction in the incidence of VAP.

DETAILED DESCRIPTION:
Patients will be enrolled following inclusion-exclusion criteria

* Base line clinical and laboratory data will be recorded in a pre designed proforma.
* Endotracheal aspirate will be taken at the time of enrollment and day3, day5, day7 and then weekly till patient is on mechanical ventilation.

Data collection

For each patient following data will be recorded as per the proforma.

During Hospitalization

All eligible patients will be carefully followed up for signs of VAP during hospitalization.

Apart from clinical examination, regular recording of body temperature, observance of tracheal aspirate appearance, leukocyte counts and chest radiograph will be done.

VAP Diagnosis: Based on American College of Chest Physicians (ACCP) criteria:

An association of a new or progressive consolidation on chest radiograph Plus at least two of the following variables

* fever > 38 degree
* leucocytosis ( > 12000) or leucopenia ( <4000)
* purulent secretions

At VAP Diagnosis

Patients who diagnosed as cases VAP, based on the above criteria.

Non-bronchoscopic bronchoalveolar lavage (BAL) will be done for microbiological sampling. In patients where clinically indicated, Flexible bronchoscopy and Bronchoalveolar lavage, sampling will be done. At the time of VAP diagnosis blood culture and urine culture, will also be sent.

Sample Collection

Endotracheal aspiration

A sterile 22 inch, 12 French suction catheter with a mucus extractor will be introduced at least 30 cm and minimum of 5ml sample will be collected. Endotracheal aspirate cultures will be examined semi quantitatively. Bacterial and antibiotic susceptibility tests will be performed.

Non bronchoscopic protected BAL

Specimen will be collected by sputum suction trap. A 47-48 cm sterile suction catheter of 16fr will be inserted through endotracheal tube till it meets resistance and will be wedged there.Then a 50cm long 8fr sterile suction catheter will be passed through it till it meets resistance and specimen will be taken. 20ml of NS instilled, minimum of 5ml aspirate will be collected. If aspirate is less than 5 ml it will be repeated.

Bronchoscopic BAL

Consent will be taken from the legal guardian. The patient will receive adequate sedation; short-acting paralytic agent to prevent coughing during the procedure Will be considered if necessary. The endotracheal tube will be ≥ 1.5 mm larger than the external diameter of the flexible bronchoscope. The patients will receive a fraction of inspired oxygen (FiO2) of 100%, and positive-end expiratory pressure will be reduced as much as tolerated. To maximize ventilation and minimize air trapping, the peak inspiratory flow will be decreased to ≤60 liters/min, the respiratory rate set between 10 and 20 breaths/ min, and the peak inspiratory pressure alarm increased. The patient will be carefully monitored throughout the procedure. The sampling area will be chosen based on the location of the infiltrate on chest X-ray.

Microbiological analysis

All the samples were subjected to Gram staining and microscopic examination and were cultured on sheep blood agar, chocolate agar and MacConkey agar semi quantitatively and 104/ml CFU was considered significant. Isolated strains were identified by standard microbiological techniques and the antimicrobial susceptibility testing were performed by disc diffusion method as per CLSI guidelines. The Gram negative bacilli were tested against the following antibiotics:amikacin, amoxicillin-clavulanate, cefotaxime, ceftazidime, ciprofloxacin, cefaperazone-sulbactam, meropenem ,imipenem, netilimicin, Piperacillin-tazobactum. Additionally colistin and ertapenem will be tested when appropriate. Gram positive organisms will be tested for amikacin, netilmicin, cotrimoxazole, ceftazidime, ciprofloxacin,cefoperazone-sulbactam, penicillin, linezolid, erythromycin, vancomycin and teicoplanin

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Requiring orotracheal intubation and mechanical ventilation

Exclusion Criteria:

* Patients intubated outside the hospital
* Patient extubated within 72 hours
* Patient already on tracheostomy
* Death occurring within 72 hours
* Pneumonia developing within 48 hours
* Patient/relatives not giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-16 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Ventilator Associated Pneumonia | 28 days
  To assess the role of endotracheal tube with subglottic suction drainage on incidence of VAP as compared to standard ET tube
Incidence of airway colonization | 28 days
  Assess the incidence of airway colonization during the period of endotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Vijay N Nongpiur, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Department of Pulmonary Medicine and Sleep Disorders, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No